CLINICAL TRIAL: NCT00891683
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of AEG33773 Versus Placebo in Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy of AEG33773 Versus Placebo in Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEG33773-201
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Diabetic Peripheral Neuropathy; Chronic Pain
Keywords: Diabetic; peripheral; neuropathy; pain; hyperalgesia; allodynia
MeSH Terms: conditions — Chronic Pain; Pain; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): 4 Capsules of Placebo
  Interventions: Drug: AEG33773 oral dosing
- 100 mg (Active Comparator): One 100 mg capsule and 3 placebo capsules of AEG33773
  Interventions: Drug: AEG33773 oral dosing
- 200 mg (Active Comparator): Two 100 mg capsules and two placebo capsules
  Interventions: Drug: AEG33773 oral dosing
- 400 mg (Active Comparator): Four 100 mg AEG33773 capsules
  Interventions: Drug: AEG33773 oral dosing

INTERVENTIONS:
Drug: AEG33773 oral dosing — AEG33773 capsules: subjects will receive a daily dose of either 100 mg, 200 mg, or 400 mg AEG33773. Placebo capsules: subjects will receive a daily dose of placebo (matching test product). Capsules will be taken by mouth, over 28 consecutive days

SUMMARY:
Two Phase 1 studies have been conducted with AEG33773 and available safety and tolerability data from these studies support further clinical development of AEG33773. The current study is proposed as a proof-of-concept study to assess the potential analgesic efficacy of AEG33773 to reduce pain associated with chronic Diabetic Peripheral Neuropathy.

DETAILED DESCRIPTION:
Doses of AEG33773 selected for evaluation in this study provide a dose range (i.e., 100-400 mg) that may potentially include both a minimally effective dose and a maximum tolerated dose. Doses up to 400 mg were well tolerated in single- and multiple-dose Phase 1 studies.

Before initiation of treatment with study drug, other analgesic medications will be discontinued during a 7-day Washout Period, and neuropathic pain will be assessed (in the absence of analgesic medication) over the next 3 days (Pain Assessment Period). Pain intensity level during these 3 days will be recorded daily, and only those subjects who meet predefined pain intensity threshold criteria on all 3 days will be eligible to receive study drug. Because pain may increase after analgesic medications have been discontinued, the combined length of the Washout and Pain Assessment Periods is limited in order that subjects who experience increased pain during this time may begin treatment with study drug without undue delay. This design will allow for adequate Baseline pain assessment over 3 days while avoiding a more prolonged period of increasing pain in the absence of analgesic medications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 75 years
* Patients with type 1 or type 2 diabetes mellitus
* DPN as determined by the investigator based on clinical history, clinical examination, and assessment of signs and symptoms
* Stable diabetic control over the preceding 3 months, as determined by the investigator based on available medical information (e.g., hemoglobin A1c [HbA1c] and/or blood glucose levels)
* HbA1c ≤ 12 % at the Screening visit
* Pain persisting for more than 3 months and less than 5 years
* Completion of 3 daily pain intensity reports (using the 11-point NPRS) over the 3 days immediately preceding the day of randomization
* Pain intensity (NPRS) score of ≥ 5 for all 3 of the 3 days immediately preceding the day of randomization
* Completed a washout (before first NPRS assessment) of at least 7 days for any of the following medications: α2-δ antagonists (e.g., gabapentin, pregabalin), opiate analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), topical lidocaine, anti-epileptic drugs, serotonin and norepinephrine reuptake inhibitors (SNRIs) (e.g., duloxetine), tricyclic antidepressants prescribed for pain, skeletal muscle relaxants, orally administered steroids, capsaicin, mexiletene, centrally acting analgesics (dextromethorphan, tramadol), alpha lipoic acid, and any supplement or herbal product used to treat DPN symptoms
* Women must be neither pregnant nor lactating. Women of childbearing age must have a confirmed negative pregnancy test and must practice medically acceptable methods of contraception throughout the trial and for at least 30 days after the last dose of study drug
* Male subjects and/or their female partners must be using medically acceptable methods of contraception for the entire duration of the study, and for at least 90 days after the last study drug dose
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* A willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Age younger than 18 years or older than 75 years
* Are pregnant or breast feeding
* Female patients of childbearing potential unwilling to use a medically acceptable form of contraception (i.e., hormonal birth control, intrauterine device [IUD], double barrier [male condom or female condom with a diaphragm], or a barrier method plus a spermicidal agent [contraceptive foam, jelly, or cream]) Female patients are considered to be of childbearing potential unless they have been postmenopausal for at least 1 year, are biologically sterile, or are surgically sterile (history of hysterectomy, bilateral oophorectomy, or bilateral tubal ligation.
* Male patients (and/or their female partners) unwilling to use a medically acceptable form of contraception during participation in the study and for at least 90 days after the last dose of study drug. Medically acceptable forms of contraception are hormonal birth control, intrauterine device (IUD), double barrier (male condom or female condom with a diaphragm), or a barrier method plus a spermicidal agent (contraceptive foam, jelly, or cream)
* Treatment with local anesthetic nerve blocks within the last 30 days before the Screening visit
* Other severe pain which may impair the self-assessment of pain due to DPN
* Participation in another study within 30 days before the Screening visit and/or during study participation
* History of drug or alcohol abuse within the past 2 years
* Creatinine clearance < 50 mL/min at the Screening visit
* Malignancy other than basal cell carcinoma and carcinoma in situ within the past 2 years
* History of chronic hepatitis B or C, hepatitis within the past 3 months before the Screening visit, or any history of human immunodeficiency virus (HIV) infection
* Clinically significant hepatic, respiratory, hematological, cardiovascular, renal, or neurological disease, with the exception of diabetic peripheral neuropathy
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times higher than the upper limit of the laboratory normal reference range at the Screening visit
* ECG with a QTcB > 470 ms at the Screening visit or at Baseline (if at either the Screening visit or Baseline the ECG shows a QTcB > 470 ms, then the investigator may immediately repeat the ECG twice and the QTcB value for inclusion/exclusion purposes will be determined by calculating the average of the 3 readings)
* Immunocompromised state
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential efficacy of AEG33773 in reducing chronic pain due to DPN | 1 year

SECONDARY OUTCOMES:
To evaluate a range of AEG33773 doses that provide efficacy | 1 year
To determine a minimally effective dose of AEG33773 | 1 year
To determine a maximally tolerated dose of AEG33773 | 1 year
To evaluate the safety and tolerability of AEG33773 | 1 year
To explore AEG33773-dependent pharmacodynamic (PD) effects in blood of patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Jolivet, MD, FRCP(C), Study Director — Aegera Therapeutics, Inc
Locations (20):
- United States (5):
  - Neurological Research Institute, Santa Monica, California
  - Radiant Research, Cincinnatti, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - Internal Department, Byala
  - University Multiprofile Hospital for Active Treatment - Clinic of Endocrinology and Metabolic Diseases, Pleven
  - University Multiprofile Hospital for Active Treatment - Clinic of Endocrinology and Metabolic Diseases, Plovdiv
  - Multiprofile Hospital for Active Treatment - Therapeutical and Endocrinology Department, Rousse
  - University Multiprofile Hospital Treatment Stara Zagora, Stara Zagora
- Canada (3):
  - Clinique d'Endocrinologie de l'Outaouais, Hull, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Hopital de l'Enfant Jesus, Québec, Quebec
- Romania (7):
  - Medical Center "Dr. Negrisanu" SRL, Timișoara, Transylvania
  - S.C. Nicodiab SRL, Bucharest
  - National Clinical Institute of Diabetes, Nutrition and Metabolic Diseases, Bucharest
  - National Institute of Diabetes Nutrition and Metabolic Diseases, Bucharest
  - Mosilor Diabetes Mellitus and Obesity Medical, Bucharest
  - Emergency Clinical County Hospital Cluj County, Cluj-Napoca
  - St. Spiridon Emergency Clinical County Hospital, Iași